CLINICAL TRIAL: NCT07202689
Title: The Predictive Value of Multimodal Brain Monitoring for Perioperative Stroke in Cardiac Surgery Patients: A Prospective Observational Study
Brief Title: The Predictive Value of Multimodal Brain Monitoring for Perioperative Stroke in Cardiac Surgery Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yuming Peng, Deputy chief of Department of Anesthesiology, Beijing Tiantan Hospital
Other Study IDs: 2025-09-10
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Multimodal Monitoring; Perioperative Stroke; Covert Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- With stroke
  Interventions: Device: Multimodal monitoring
- Without stroke
  Interventions: Device: Multimodal monitoring

INTERVENTIONS:
Device: Multimodal monitoring — Multimodal monitoring technology offers a novel approach to cerebral protection during the perioperative period of cardiac surgery by integrating hemodynamic parameters, autonomic nervous responses, cerebral oxygen saturation and indices, electroencephalographic activity, and cerebral blood flow velocity.

SUMMARY:
Postoperative stroke following cardiac surgery is associated with a ninefold increase in mortality risk compared to patients without stroke. Perioperative monitoring in cardiac surgery involves a range of complex and diverse techniques, presenting significant challenges for anesthetic management. Multimodal brain monitoring technology offers a novel approach to cerebral protection during the perioperative period of cardiac surgery by integrating hemodynamic parameters, autonomic nervous responses, cerebral oxygen saturation and indices, electroencephalographic activity, and cerebral blood flow velocity. Therefore, this study aims to evaluate the comprehensive early-warning efficacy of multimodal brain monitoring for perioperative stroke in cardiac surgery patients, determine the cumulative incidence of perioperative stroke-including covert stroke-and provide a new theoretical basis for optimizing cerebral protection strategies in cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective cardiac surgery
* Presence of at least one of the following high-risk factors for stroke: a.Peripheral vascular disease (history of peripheral artery bypass grafting, amputation for ischemia, Ankle-Brachial Pressure Index < 0.9, or history of abdominal aortic aneurysm repair).b.Cerebrovascular disease (history of stroke, transient ischemic attack, or carotid stenosis >70%).c.Renal insufficiency (Glomerular Filtration Rate < 60 mL/min/1.73m²).d.Diabetes mellitus (requiring oral hypoglycemic agents and/or insulin therapy).e.Urgent coronary artery bypass grafting (inpatient requiring revascularization due to acute coronary syndrome or myocardial infarction).f.Recent smoking history (within 1 year).g.Left ventricular ejection fraction < 35%
* Provision of signed informed consent

Exclusion Criteria:

* Contraindication to magnetic resonance imaging (e.g., claustrophobia, inability to lie flat for the duration of the study, presence of a pacemaker or implantable cardioverter-defibrillator, or other metallic implants)
* Inability to complete cognitive function assessments
* Patients with psychiatric, legal disabilities or under legal guardianship
* Life expectancy of less than 3 months
* Women who are lactating or pregnant
* Diagnosis of any type of dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population will be selected from patients who schedule to receive elective cardiac surgery in Beijing Tiantan Hospital.
Sampling Method: Probability Sample
Enrollment: 369 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of perioperative stroke | 48 hours preoperatively and 3-7 days postoperatively
  Perioperative stroke is diagnosed by MRI

CONTACTS AND LOCATIONS:
Overall Officials: Yuming Peng, MD,Ph.D, Principal Investigator — Beijing Tiantan Hospital

IPD SHARING:
Plan to Share IPD: No